CLINICAL TRIAL: NCT05557500
Title: Assessment of Psychological Symptoms and Quality if Life Among Fibromyalgia Patients and Its Risk Factors
Brief Title: Assessment of Psychological Symptoms Among Fibromyalgia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, CA Adeeb, Principal investigator, Assiut University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: APF
Record Dates: First submitted 2022-09-25; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Psychological Symptoms in Fibromyalgia Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibromyalgia patients with use of rtms sessions for treatment (Experimental): Repitetive transcranial magnetic stimulation on primary motor area with 20 HZ for 20 sessions
  Interventions: Device: Repitetive transcranial magnetic stimulation
- Fibromyalgia pt with use of sphenopalatine ganglion block as treatment (Experimental): Pain killing intervention for pain control of myofacial pain in fibromyalgia patients
  Interventions: Device: Repitetive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repitetive transcranial magnetic stimulation — Repitetive transcranial magnetic stimulation on primary motor area with 20 HZ for 20 sessions

SUMMARY:
Fibromyalgia is a syndrome characterized by chronic widespread pain at multiple tender points, joint stiffness, and systemic symptoms (e.g., mood disorders, fatigue, cognitive dysfunction, and insomnia) [14] without a well-defined underlying organic disease. Nevertheless, it can be associated with specific diseases such as rheumatic pathologies, psychiatric or neurological disorders, infections, and diabetes.

The prevalence of fibromyalgia has been estimated to be around 1%-2% (3.4% for women and 0.5% for men) [5, 6].

DETAILED DESCRIPTION:
The etiology and pathogenesis of fibromyalgia are still not fully understood. Several factors such as dysfunction of the central and autonomic nervous systems, neurotransmitters, hormones, immune system, external stressors, psychiatric aspects, and others seem to be involved.

diagnosis is principally based on the two major diagnostic criteria defined by the ACR in 1990 [7]: (1) a history of widespread musculoskeletal pain present for at least three months, and (2) tenderness in at least 11 of 18 defined tender points

Psychiatric problems seem to contribute considerably to the development of fibromyalgia. The prevalence of psychiatric conditions among patients affected by fibromyalgia is higher than among subjects complaining of other rheumatic diseases . The most common disorders associated are anxiety, somatization, dysthymia, panic disorders, posttraumatic stress, and overall depression [8]. Depression is more frequently associated with fibromyalgia than with other musculoskeletal diseases [9] Depression worsens fibromyalgic symptoms and vice versa, and antidepressants represent a cornerstone of fibromyalgia therapy [1011].

Over the last decade, it has been repeatedly shown that noninvasive repetitive transcranial magnetic stimulation (rTMS) of the primary motor cortex (M1) induces analgesic effects both in experimental pain [1216] , probably by activating pain modulation systems.

Another way studied to relieve fibromyalgia pain is sphenopalatine ganglion block

In our study we will evaluate the effect of repetitive transcranial magnetic stimulation and sphenopalatine ganglion block on fibromyalgia pain and psychiatric symptoms.

rtms will be applied on primary motor area (M1) for 20 sessions (5 daily per week for 4 weeks)with 20 HZ and 3000pul with evaluation of pain and psychological symptoms befor intervention and after 10 sesions and after 1 month of last session compared to sphenopalatine ganglion block effect .

ELIGIBILITY:
Inclusion Criteria:

- Women aged from 18 to 60 years old Diagnosed as fibromyalgia with resistence to pharmacological treatment

Exclusion Criteria:

* Previous psychiatric disorders Sever cognitive dysfunction Other medical or neurological disorders Pregnant females

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate prevelance of psychiatric disorders among fibromyalgia patients | 3 years
  Identify possible risk factors that lead to psychiatric illness in fibromyalgia patients Evaluate effect of non pharmacological treatment in form of sphenopalatine ganglion block and transcranial mag netic stimulation on psychiatric symptoms in fibromyalgia patients

REFERENCES:
- [Background] Bigatti SM, Hernandez AM, Cronan TA, Rand KL. Sleep disturbances in fibromyalgia syndrome: relationship to pain and depression. Arthritis Rheum. 2008 Jul 15;59(7):961-7. doi: 10.1002/art.23828. PMID 18576297
- [Background] Clauw DJ. Fibromyalgia: a clinical review. JAMA. 2014 Apr 16;311(15):1547-55. doi: 10.1001/jama.2014.3266. PMID 24737367
- [Background] Giesecke T, Williams DA, Harris RE, Cupps TR, Tian X, Tian TX, Gracely RH, Clauw DJ. Subgrouping of fibromyalgia patients on the basis of pressure-pain thresholds and psychological factors. Arthritis Rheum. 2003 Oct;48(10):2916-22. doi: 10.1002/art.11272. PMID 14558098
- [Background] Mease P. Fibromyalgia syndrome: review of clinical presentation, pathogenesis, outcome measures, and treatment. J Rheumatol Suppl. 2005 Aug;75:6-21. PMID 16078356
- [Background] Wolfe F, Ross K, Anderson J, Russell IJ, Hebert L. The prevalence and characteristics of fibromyalgia in the general population. Arthritis Rheum. 1995 Jan;38(1):19-28. doi: 10.1002/art.1780380104. PMID 7818567
- [Background] Lindell L, Bergman S, Petersson IF, Jacobsson LT, Herrstrom P. Prevalence of fibromyalgia and chronic widespread pain. Scand J Prim Health Care. 2000 Sep;18(3):149-53. doi: 10.1080/028134300453340. PMID 11097099
- [Background] Sarzi-Puttini P, Atzeni F, Di Franco M, Lama N, Batticciotto A, Iannuccelli C, Dell'Acqua D, de Portu S, Riccieri V, Carrabba M, Buskila D, Doria A, Valesini G. Anti-polymer antibodies are correlated with pain and fatigue severity in patients with fibromyalgia syndrome. Autoimmunity. 2008 Feb;41(1):74-9. doi: 10.1080/08916930701620035. PMID 18176867
- [Background] Katon W, Sullivan M, Walker E. Medical symptoms without identified pathology: relationship to psychiatric disorders, childhood and adult trauma, and personality traits. Ann Intern Med. 2001 May 1;134(9 Pt 2):917-25. doi: 10.7326/0003-4819-134-9_part_2-200105011-00017. PMID 11346329
- [Background] [1990 classification criteria of fibromyalgia from the American College of Rheumatology. Report of the Multicenter Criteria Committee]. Union Med Can. 1990 Sep-Oct;119(5):272. No abstract available. French. PMID 2238278
- [Background] Andre-Obadia N, Peyron R, Mertens P, Mauguiere F, Laurent B, Garcia-Larrea L. Transcranial magnetic stimulation for pain control. Double-blind study of different frequencies against placebo, and correlation with motor cortex stimulation efficacy. Clin Neurophysiol. 2006 Jul;117(7):1536-44. doi: 10.1016/j.clinph.2006.03.025. Epub 2006 Jun 5. PMID 16753335
- [Background] Graff-Guerrero A, Gonzalez-Olvera J, Fresan A, Gomez-Martin D, Mendez-Nunez JC, Pellicer F. Repetitive transcranial magnetic stimulation of dorsolateral prefrontal cortex increases tolerance to human experimental pain. Brain Res Cogn Brain Res. 2005 Sep;25(1):153-60. doi: 10.1016/j.cogbrainres.2005.05.002. PMID 15935625
- [Background] Summers J, Johnson S, Pridmore S, Oberoi G. Changes to cold detection and pain thresholds following low and high frequency transcranial magnetic stimulation of the motor cortex. Neurosci Lett. 2004 Sep 23;368(2):197-200. doi: 10.1016/j.neulet.2004.07.008. PMID 15351448
- [Background] Valmunen T, Pertovaara A, Taiminen T, Virtanen A, Parkkola R, Jaaskelainen SK. Modulation of facial sensitivity by navigated rTMS in healthy subjects. Pain. 2009 Mar;142(1-2):149-58. doi: 10.1016/j.pain.2008.12.031. Epub 2009 Feb 6. PMID 19201092
- [Background] Nahmias F, Debes C, de Andrade DC, Mhalla A, Bouhassira D. Diffuse analgesic effects of unilateral repetitive transcranial magnetic stimulation (rTMS) in healthy volunteers. Pain. 2009 Dec 15;147(1-3):224-32. doi: 10.1016/j.pain.2009.09.016. Epub 2009 Oct 12. PMID 19822394